CLINICAL TRIAL: NCT01154153
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating the Pharmacodynamic Effect of a 6-week Treatment With Triamcinolone Acetonide Aqueous Nasal Spray 110 μg and 220 μg Once Daily on Basal Hypothalamic-Pituitary-Adrenal (HPA) Axis Function in Children [>=2 to < 12 Years of Age] With Allergic Rhinitis (AR).
Brief Title: Nasacort AQ Hypothalamic-Pituitary-Adrenal (HPA) Axis Study in Children With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRICA_L_04286
Record Dates: First submitted 2010-06-22; First posted 2010-06-30 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Rhinitis, Allergic, Perennial and/or Seasonal
MeSH Terms: conditions — Rhinitis | interventions — Nasal Sprays; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): * placebo during the screening phase and
  * placebo during the treatment phase.
  All children had the option to take rescue medication, (Claritin®) as needed to relieve symptoms of AR.
  Interventions: Drug: Placebo nasal spray; Drug: Claritin® Syrup
- TAA-AQ (Experimental): * placebo during the screening phase and
  * TAA-AQ (Nasacort AQ) during the treatment phase.
  All children had the option to take rescue medication, (Claritin®) as needed to relieve symptoms of AR.
  Interventions: Drug: Placebo nasal spray; Drug: Triamcinolone acetonide aqueous (TAA-AQ) nasal spray (NASACORT AQ); Drug: Claritin® Syrup

INTERVENTIONS:
Drug: Placebo nasal spray — 1 spray/nostril, once daily in the morning, for 8 to 24 days during the screening phase.
Drug: Triamcinolone acetonide aqueous (TAA-AQ) nasal spray (NASACORT AQ) — Treatment assignment was randomized with stratification by sex and age group (>=2 to <6, >=6 to <12 years old).
  * For children who were >=2 to <6 years old, 1 spray/nostril (110 µg TAA-AQ), once daily in the morning, for 6 weeks, during the double-blind treatment phase.
  * For children who were >=6 yrs to <12 years old, either 1 spray/nostril (110 µg TAA-AQ) or 2 sprays/nostril (220 µg TAA-AQ), once daily in the morning, for 6 weeks, during the double-blind treatment phase.
  Arms: TAA-AQ
Drug: Placebo nasal spray — Treatment assignment was randomized with stratification by sex and age group (>=2 to <6, >=6 to <12 years old).
  * For children who were >=2 to <6 years old, 1 spray/nostril, once daily in the morning, for 6 weeks, during the double-blind treatment phase.
  * For children who were >= 6 yrs to <12 years old, either 1 spray/nostril or 2 sprays/nostril, once daily in the morning, for 6 weeks, during the double-blind treatment phase.
  Arms: Placebo
Drug: Claritin® Syrup — Children's Claritin® Syrup [5 mg of loratadine per 5 mL] could be taken orally for the relief of AR symptoms throughout the study on an as needed basis, according to the Food and Drug Administration-approved manufacturer's label.

SUMMARY:
The primary objective was to evaluate the effect of a 6-week treatment with TAA-AQ (110 μg) and TAA-AQ (220 μg) once daily (QD) versus placebo on hypothalamic-pituitary-adrenal (HPA) axis function as measured by serum cortisol AUC(0-24 hr) in children (>=2 to <12 years old) with allergic rhinitis (AR).

DETAILED DESCRIPTION:
The study consisted of a run-in single-blind screening phase (prerandomization) followed by an approximately 6-week double-blind treatment phase (postrandomization).

Total study duration per participant lasted from 7.5 to 13 weeks and consisted of:

* Screening and single-blind phases (these 2 phases ran concurrently, prerandomization) for 8 to 24 days. During the screening phase participants were given a single-blind placebo nasal spray to enable them to practice their intranasal application technique once daily in the morning (1 actuation/nostril).
* Randomization to the double-blind treatment phase. Treatment assignment was randomized with stratification by sex and age group (>=2 to <6, >=6 to <12 years old).
* Double-blind treatment phase which lasted at least 42 days and ran up to 47 days. Participants were administered either TAA-AQ nasal spray or placebo nasal spray.
* An evaluation at the end of treatment 1-3 days after completion of the double-blind phase.

ELIGIBILITY:
Participants who met the following criteria were eligible for this study:

Inclusion Criteria:

* History of AR documented by the investigator, as follows:

  * At least a 1-year clinical history (6-month history if the participant was >= 2 to < 4 years of age) of perennial allergic rhinitis (PAR); or a clinical history of seasonal allergic rhinitis (SAR) over 2 seasons and
  * positive skin test (prick or intradermal) to a seasonal or perennial allergen that was present in the participant's environment at time of screening.
* Written informed consent and ability of parent/legal guardian of the participant to give a written informed consent before any study related procedures. Participants >=7 years of age (or younger according to the governing institutional review board [IRB]) had to provide a signed assent form

Exclusion Criteria:

* Concomitant medical condition that might have interfered with the administration of a nasal spray, including anatomical abnormalities of the nose, face (eg, polyposis, markedly deviated septum)
* Presence of any active, untreated, or clinically significant musculoskeletal, endocrinologic, gastrointestinal, hepatic, respiratory, cardiovascular, or neurological condition that might have interfered with the study
* Any conditions or treatment that might have affected the HPA axis or the plasma cortisol assay, including but not limited to:

  * Documented disorder involving the hypothalamus, pituitary, or adrenal gland
  * Current use of serotonergic, dopaminergic, adrenergic, cholinergic agonists and antagonists, opiates, immunomodulatory, hormonal drugs, and lipid-lowering agents
  * Treatment with systemic corticosteroids (oral, intravenous, intramuscular, or intra-articular) within 3 months prior to Visit 1
  * Treatment with systemic corticosteroids for > 2 courses received up to 1 year before Visit 1 was exclusionary. Up to 2 courses of systemic corticosteroids, each course not exceeding 14 days, up to 1 year before Visit 1 was allowed
  * Treatment with inhaled, intranasal, or high-potency topical corticosteroids within 6 weeks of Visit 1
  * History of hospitalization due to asthma within 1 year before screening. Participants with mild asthma that was well-controlled without the use of inhaled corticosteroids within 6 weeks prior to Visit 1 were eligible for the study
* Any clinically significant (as determined by the investigator) abnormal laboratory test at Visit 1
* Morning serum cortisol outside the reference range at Visit 1
* Any of the following missing serum cortisol samples from the Visit-2 collection: first sample (before administration of investigational product), 20-hour sample, 24-hour sample, or any 2 consecutive samples
* Any medical condition where use of corticosteroids might have been contraindicated or could have led to disease exacerbation (eg, glaucoma, cataract, ocular herpes simplex, tuberculosis, growth retardation)
* History of hypersensitivity to corticosteroids or to the rescue medication, investigational product, or to any of their excipients
* Unresolved upper respiratory tract infection, sinus infection, or nasal candidiasis (ie, symptomatic or under treatment) within the last 2 weeks prior to Visit 1 and Visit 3
* Females of childbearing potential not protected by effective contraceptive method of birth control or were unwilling to abstain from sexual activity and/or, were unwilling or unable to test for pregnancy. Only female adolescent with onset of menses were to be checked by serum pregnancy test at Visit 1
* Pregnant female adolescent (who tested positive for pregnancy at Visit 1) The above information was not intended to contain all considerations relevant to potential participation in a clinical trial.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (8):
- United States (8):
  - Investigational Site Number 840003, Cypress, California
  - Investigational Site Number 840006, Stockbridge, Georgia
  - Investigational Site Number 840007, North Dartmouth, Massachusetts
  - Investigational Site Number 840010, Plymouth, Minnesota
  - Investigational Site Number 840001, Omaha, Nebraska
  - Investigational Site Number 840008, Raleigh, North Carolina
  - Investigational Site Number 840002, Spartanburg, South Carolina
  - Investigational Site Number 840005, San Antonio, Texas

REFERENCES:
- [Derived] Georges G, Kim KT, Ratner P, Segall N, Qiu C. Effect of intranasal triamcinolone acetonide on basal hypothalamic-pituitary-adrenal axis function in children with allergic rhinitis. Allergy Asthma Proc. 2014 Mar-Apr;35(2):163-70. doi: 10.2500/aap.2014.35.3728. PMID 24717794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in 8 study centers in the United States.
Pre-assignment Details: 179 participants were screened in this study. 31 participants were screen failures and 8 participants did not continue to as the limit on the number of participants to be randomized had been reached. 140 participants were randomized.
Groups:
- Placebo: Children >=2 to <12 years old with AR symptoms who received placebo during the screening phase and placebo during the treatment phase. All children had the option to take rescue medication, (Claritin®) as needed to relieve symptoms of AR.
- TAA-AQ: Children >=2 to <12 years old with AR symptoms who received placebo during the screening phase and TAA-AQ (Nasacort AQ) during the treatment phase. All children had the option to take rescue medication, (Claritin®) as needed to relieve symptoms of AR.
Period: Overall Study
Arm/Group | Placebo | TAA-AQ
Started | 71 | 69
Completed | 66 | 66
Not Completed | 5 | 3
Not completed — Poor compliance to protocol | 2 | 0
Not completed — Unable to use labs | 2 | 3
Not completed — Withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAA-AQ | Total
Number analyzed (Participants) | 71 | 69 | 140
Age Continuous [Mean (Standard Deviation); unit: years] | 7.3 (2.7) | 7.1 (2.5) | 7.2 (2.6)
Age, Customized [Number; unit: participants]
  >=2 to < 4 years | 6 | 5 | 11
  >=4 to < 6 years | 15 | 16 | 31
  >=6 to < 12 years | 50 | 48 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 42 | 41 | 83
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 43 | 42 | 85
  Others | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 71 | 69 | 140
Tanner Classification [Number; unit: Participants] — Tanner classification distinguishes stages of puberty. Each stage represents the extent of breast, genitalia and pubic hair growth. Tanner Stage I represents the pre-adolescent stage where breast, genitalia and pubic hair growth are of the same size and shape as in early childhood and in Tanner Stage 5 breasts and genitalia are of adult shape and size, and pubic hair is adult in quantity (mature stage). Stages 2, 3 and 4 are intermediate stages.
  Participants
    Stage 1 | 55 | 60 | 115
    Stage 2 | 12 | 9 | 21
    Stage 3 | 4 | 0 | 4
    Stage 4 | 0 | 0 | 0
    Stage 5 | 0 | 0 | 0
Primary Allergic Rhinitis (AR) diagnosis [Number; unit: Participants] — Participants diagnosed with perennial allergic rhinitis (PAR); and seasonal allergic rhinitis (SAR).
  Participants
    PAR only | 11 | 12 | 23
    SAR only | 5 | 3 | 8
    Both PAR and SAR | 55 | 54 | 109
Time from the first Allergic Rhinitis symptom to Visit 1 [Mean (Standard Deviation); unit: Years] — For participants with both PAR and SAR, it is the longest time. A missing month of the first symptom start date was imputed as December and a missing day was imputed as the last date of the month.
  Years | 4.82 (2.70) | 4.79 (2.48) | 4.80 (2.59)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Serum Cortisol Area Under Curve [AUC(0-24 hr)] at the End of Treatment to Baseline
Description: Blood samples were collected over a 24-hour period (at 0, 2, 4, 8, 12, 20, and 24 hours), with 0 hour being between 8:00AM to 9:00AM, immediately prior to investigational product (IP) administration. AUC (0-24hr) was calculated using the trapezoid rule, and was normalized by dividing the AUC(0-24 hr) by the actual sample collection interval between 0-hour and 24-hour blood draw times.
  Ratio in Serum Cortisol AUC(0-24 hr) = (Serum Cortisol AUC[0-24 hr] at 6 weeks postrandomization)/(Serum Cortisol AUC[0-24 hr] at 1-3 days prerandomization). Log transformation was used for the analysis.
Time Frame: 1-3 days prerandomization and 6 weeks postrandomization
Population: The per protocol (PP) population included all randomized participants who took at least one dose of study medication and had no major protocol violations. Major protocol violations were those deemed most likely to affect the interpretation of the results and included poor compliance, use of prohibited medication, missing blood samples.
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Ratio | 0.938 [0.39 to 1.63] | 0.898 [0.48 to 4.45]
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Missing cortisol values were imputed with multiple imputation. AUC(0-24 hr) was calculated for each imputation and analyzed with log-transformation using an ANCOVA model and analyzed with treatment, sex, and age group as fixed effects, and log-transformed baseline value as a covariate. The mean difference in log scale between treatments and its standard error were calculated by Least Squares mean. Results from multiply imputed data were combined using SAS procedure MIANALYZE; Test type: Superiority or Other; ANCOVA; Treatment Ratio of Geometric mean = 0.966, 95% CI 2-sided [0.892 to 1.045] — The treatment ratio was calculated as an exponential of the mean difference between treatments in log scale

2. Secondary Outcome: Change From Baseline in the Reflective Total Nasal Symptom Score (rTNSS)
Description: Every morning, participants rated the severity of symptoms experienced over the previous 24 hours using scale from 0-3, where 0=symptoms absent, 1=mild, 2=moderate, and 3=severe symptoms (interfere with daily living or sleep) for each symptom (nasal congestion, nasal itching, sneezing, and runny nose). The rTNSS was the sum of the individual symptom scores, ranged from 0-12 (where 12 reflected the worst symptoms).
  Change from baseline in the rTNSS = mean rTNSS (double-blind treatment phase) - mean rTNSS (screening phase).
Time Frame: From 8-24 days prerandomization up to 6 weeks postrandomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Score on a scale | -0.22 (1.12) | -1.07 (1.66)
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Test type: Superiority or Other; p = 0.0007, ANCOVA; For ANCOVA, treatment arm, randomization strata were fixed effects and baseline value was a covariate; LS Mean Difference = -0.85, 95% CI 2-sided [-1.34 to -0.37], Standard Error of Mean 0.24

3. Secondary Outcome: Number of Participants by Relief Level as Evaluated by the Physician
Description: Efficacy of treatment was assessed by the physician using a scale from 0-4 for relief levels, where 0 = no relief (symptoms unchanged or worsened than before), 1 = slight relief (symptoms present and only minimally improved), 2 = moderate relief (symptoms are present and may be troublesome, but are noticeably improved), 3 = marked relief (symptoms are greatly improved and although present are scarcely troublesome) and 4 = complete relief (virtually no symptom present).
Time Frame: At end of study (43-50 days after randomization)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Participants
  Relief Level 0 (No relief) | 11 | 9
  Relief Level 1 (Slight relief) | 18 | 13
  Relief Level 2 (Moderate relief) | 16 | 20
  Relief Level 3 (Marked relief) | 13 | 17
  Relief Level 4 (Complete relief) | 3 | 6
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Test type: Superiority or Other; p = 0.1332, Cochran-Mantel-Haenszel — Based on the ordinal evaluation score and adjusted for the randomization strata

4. Secondary Outcome: Number of Participants by Relief Level as Evaluated by the Participant
Description: Efficacy of treatment was assessed by the participant using a scale from 0-4 for relief levels, where 0 = no relief (symptoms unchanged or worsened than before), 1 = slight relief (symptoms present and only minimally improved), 2 = moderate relief (symptoms are present and may be troublesome, but are noticeably improved), 3 = marked relief (symptoms are greatly improved and although present are scarcely troublesome) and 4 = complete relief (virtually no symptom present).
Time Frame: At end of study (43-50 days after randomization)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Participants
  Relief level 0 (No relief) | 9 | 5
  Relief level 1 (Slight relief) | 17 | 22
  Relief level 2 (Moderate relief) | 16 | 13
  Relief level 3 (Marked relief) | 14 | 16
  Relief level 4 (Complete relief) | 5 | 9
Statistical Analysis 1: Comparison: Placebo vs TAA-AQ; Test type: Superiority or Other; p = 0.3314, Cochran-Mantel-Haenszel — Based on the ordinal evaluation score and adjusted for the randomization strata

5. Secondary Outcome: Number of Participants Using Rescue Medication
Description: The number of participants using the rescue medication (Claritin®) during the single-blind screening phase (the time from 8-24 days before randomization up to the day before randomization) and during the double-blind treatment phase (the time from randomization to end of study).
Time Frame: From 8 to 24 days prerandomization and randomization to end of study (43-50 days postrandomization)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Participants
  Prerandomization period | 8 | 8
  Postrandomization period | 24 | 19

6. Secondary Outcome: The Percent of Days of Rescue Medication Use During the Double-blind Treatment Phase
Description: The percent of days of rescue medication used during the double-blind treatment phase was calculated. For participants who did not use any rescue medication, the percentage of days using rescue medication was set to be 0.
Time Frame: From randomization to 43-50 days postrandomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo | TAA-AQ
Number analyzed (Participants) | 61 | 65
Percentage of days | 4.02 (12.77) | 3.07 (11.82)

ADVERSE EVENTS:
Arm/Group | Placebo | TAA-AQ
Serious Adverse Events (participants affected / at risk) | 1/71 | 0/69
Other Adverse Events (participants affected / at risk) | 12/71 | 7/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | TAA-AQ (N=69)
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | TAA-AQ (N=69)
Headache (Nervous system disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pyrexia (General disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication for review and comment at least 45 days (for abstracts -20 days) in advance of any submission for publication. The Sponsor may request for the publication to be delayed for a limited time, not to exceed 90 days to preserve its proprietary rights.